CLINICAL TRIAL: NCT06384560
Title: Neoadjuvant Triple Treatment with FOLFIRINOX Plus Pembrolizumab and SABR in Patients with Borderline Resectable Pancreatic Cancer (PREOPANC-5): a Multicenter Single Arm Phase I/II Trial of the Dutch Pancreatic Cancer Group
Brief Title: Neoadjuvant Triple Treatment for Borderline Resectable Pancreatic Cancer (PREOPANC-5)
Acronym: PREOPANC-5
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Maastricht University Medical Center (Other); Erasmus Medical Center (Other); St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Trial Office Medical Oncology VUmc, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508707-20-00
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Borderline Resectable Pancreatic Cancer
Keywords: borderline pancreatic cancer; neoadjuvant treatment; checkpoint inhibition; chemotherapy; stereotactic radiotherapy; surgical resection; progression free survival
MeSH Terms: interventions — pembrolizumab; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant FOLFIRINOX, SABR and pembrolizumab (Experimental): Treatment starts with four cycles of neoadjuvant FOLFIRINOX chemotherapy every two weeks, combined with pembrolizumab every six weeks, starting at the same day as the second cycle of FOLFIRINOX. Restaging is performed after cycle 4 of FOLFIRINOX with a CT-scan. Patients with a response or stable disease will undergo SABR 5 X 8 Gy followed by an additional four cycles FOLFIRNOX chemotherapy, combined with pembrolizumab. Restaging is repeated after 8 cycles FOLFRINOX in total. Patients undergo a surgical exploration if they have non-metastatic borderline resectable disease on CT-scan of the chest and abdomen, 3-6 weeks after completion of chemotherapy. Patients also proceed to surgical exploration if they discontinue neoadjuvant FOLFIRINOX and/or pembrolizumab because of toxicity or have local progression at restaging within criteria for borderline resectable disease.
  Interventions: Drug: Pembrolizumab; Drug: Folfirinox; Radiation: SABR

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 400 mg will be administered as a 30 minute IV infusion every 6 weeks.
Drug: Folfirinox — FOLFIRINOX is a combination of systemic chemotherapy agents. FOLFIRINOX consists of oxaliplatin at a dose of 85 mg/m2, given as a 2-hour intravenous infusion, immediately followed by leucovorin at a dose of 400 mg/m2 given as a 2-hour intravenous infusion, with the addition, after 30 minutes, of irinotecan at a dose of 150 mg/m2, given as a 90-minute intravenous infusion through a Y-connector. This treatment is followed by a continuous intravenous infusion of 2400 mg/m2 5-FU over a 46-hour period every 2 weeks. (The FOLFIRINOX given in the trial is the modified scheme, whereby the fluorouracil bolus at a dose of 400 mg/m2 is omitted and the irinotecan dose reduced to 150 mg/m2).
Radiation: SABR — SABR will be delivered in an image-guided hypofractionated scheme of 5 fractions of 8 Gy (total 40 Gy), prescribed to 95% of the planning target volume (PTV). Treatment is delivered on five non-consecutive days.

SUMMARY:
Since patients with borderline resectable pancreatic cancer (BRPC) have a limited life expectancy, it is important to improve treatment strategies. Therefore, the objective of this study is to investigate whether neoadjuvant triple treatment chemotherapy, immunotherapy and radiotherapy, followed by surgery and chemotherapy and immunotherapy survival in patients with BRPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic cancer
* Male or female participants who are at least 18 years of age on the day of signing in-formed consent
* Borderline resectable tumor (see table 1 for definitions of resectability)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Ability to undergo surgery, radiotherapy and chemotherapy
* Leucocytes (WBC) ≥ 3.0 X 109/l
* Platelets ≥ 100X 109 /l
* Hemoglobin ≥ 6 mmol/l
* Renal function: E-GFR > 50 ml/min
* Bilirubin < 50 µmol/l or planned for biliary drainage
* A male participant must agree to use a contraception as detailed in Appendix 5 of this protocol during the treatment period and for at least 18 weeks after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant (see Appendix 5), not breastfeeding, or a woman of childbearing potential (WOCBP) who agrees to follow the contraceptive guidance during the treatment period and for at least 18 weeks after the last dose of study treatment.
* Written informed consent

Exclusion Criteria:

* Metastatic or locally advanced (i.e. unresectable) pancreatic cancer.
* Ampullary or distal bile duct cancer.
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator.
* Complete dihydropyrimidine dehydrogenase deficiency.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to start of treatment / (see Appendix 5). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or antiPDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents for pancreatic cancer.
* Has received prior radiotherapy within 2 weeks of start of study intervention.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. COVID vaccines are allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid thera-py (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treat-ment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has cur-rent pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus infection.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* Has contra-indications for MRI (only for Amsterdam UMC and UMC Utrecht)

  * Pacemakers or implanted defibrillators, deep brain stimulators, cochlear im-plants.
  * Patients who have a metallic foreign body in their eye, or who have an aneu-rysm clip in their brain, cannot have an MRI scan since the magnetic field may dislodge the metal.
  * Patients with severe claustrophobia not able to tolerate an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with progression free survival at 18 months (RECIST 1.1) | 18 months

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Center, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No